CLINICAL TRIAL: NCT06104800
Title: Effect of Weight Loss on Hepcidin Levels and Iron Status in Subjects with Obesity.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Martha Guevara Cruz, Principal Investigator, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FNU-4686-23-24-1
Record Dates: First submitted 2023-10-18; First posted 2023-10-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Obesity; Iron Deficiency Anemia
MeSH Terms: conditions — Obesity; Anemia, Iron-Deficiency | interventions — Caloric Restriction; Red Meat

STUDY DESIGN:
Intervention Model Description: The groups will receive the treatment simultaneously.
Who Masked: Outcomes Assessor
Masking Description: The person who will perform the biochemical determinations and the statistical analysis will be blinded from the intervention group by assigning each patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Red meat diet (Experimental): Calorie-restricted diet with macronutrient distribution: 1.5 g/kg of ideal body weight in protein (including red meat), 50% carbohydrates, and 25-30% fats.
  Interventions: Other: Calorie-restricted diet with red meat
- Red meat free diet (Active Comparator): Calorie-restricted diet with macronutrient distribution: 1.5 g/kg of ideal body weight in protein (excluding red meat), 50% carbohydrates, and 25-30% fats
  Interventions: Other: Calorie-restricted diet without red meat

INTERVENTIONS:
Other: Calorie-restricted diet with red meat — Calorie-restricted diet with macronutrient distribution: 1.5 g/kg of ideal body weight in protein (including red meat), 50% carbohydrates, and 25-30% fats.
  Arms: Red meat diet
Other: Calorie-restricted diet without red meat — Calorie-restricted diet with macronutrient distribution: 1.5 g/kg of ideal body weight in protein (excluding red meat), 50% carbohydrates, and 25-30% fats
  Arms: Red meat free diet

SUMMARY:
Obesity and iron deficiency are the nutritional disorders with the highest prevalence worldwide. Different mechanisms have been proposed to explain iron deficiency secondary to obesity. Among the most studied is the deficit in dietary iron intake or the increase in blood volume that increases the need for the metal. However, one of the most plausible mechanisms linking obesity and iron deficiency is low-grade systemic inflammation, through the iron metabolism intermediate known as hepcidin. The investigators objective is to evaluate the effect of weight loss by caloric restriction on hepcidin and serum iron concentration in people living with obesity and iron deficiency. The study will be divided into two phases: Phase 1: A cross-sectional study (cases and controls) to compare hepcidin levels, iron status and inflammatory markers in people living with and without obesity. The second phase consists of an open-label randomized controlled clinical trial. Individuals living with obesity who are iron deficient will be recruited and randomized to one of 2 dietary intervention groups with 60-day follow-up. The intervention groups will be: diet with caloric restriction rich in protein (with red meat) and diet with caloric restriction rich in protein (without red meat). Hepcidin levels, iron status and inflammatory markers will be determined at the beginning and end of the intervention. The nutritional intervention will have the following distribution of macronutrients in the diet: protein 1.5 g/kg of ideal weight, 50% carbohydrates and 25-30% fats.

DETAILED DESCRIPTION:
The study will consist of two phases: Phase 1, which will be cross-sectional, and Phase 2, which will involve a randomized controlled clinical trial.

Phase 1: Cross-Sectional Study A cross-sectional study will be conducted to compare hepcidin levels, iron status and inflammatory markers in people living with and without obesity. Upon obtaining signed consent, participants will undergo a medical history assessment, anthropometric measurements (weight, height, waist circumference), body composition analysis (% body fat, % skeletal muscle mass, % fat-free mass), and blood samples will be collected to determine serum hepcidin levels, iron status, inflammatory markers (C-reactive protein, interleukin-6, lipopolysaccharides), and oxidative stress markers (MDA).

Additional blood samples will be taken for biochemical tests (glucose, lipid profile, creatinine, urea, liver function tests), insulin, leptin, adiponectin, and, optionally, DNA isolation for polymorphisms determination and those associated with iron metabolism and obesity. Participants will also complete a food frequency questionnaire (SNUT).

Phase 2: Open randomized controlled clinical trial This phase will be conducted to assess the impact of weight loss on hepcidin levels, iron status, and inflammatory markers in individuals living with obesity. Participants recruited for this phase will be selected from those identified in the first phase who exhibit iron deficiency (serum iron < 50 mcg/dL).

Participants will be randomly assigned to one of two dietary intervention groups, both of which will undergo a 60-day follow-up period with a calorie-restricted diet, reducing caloric intake by less than 25% of the resting energy expenditure determined by indirect calorimetry. The intervention groups will be as follows:

* Calorie-restricted diet with macronutrient distribution: 1.5 g/kg of ideal body weight in protein (including red meat), 50% carbohydrates, and 25-30% fats.
* Calorie-restricted diet with macronutrient distribution: 1.5 g/kg of ideal body weight in protein (excluding red meat), 50% carbohydrates, and 25-30% fats.

Additionally, all participants will receive ferrous sulfate 200mg every 48 hours for three months to correct iron-deficiency anemia.

During the initial and final visits, participants will undergo a 24-hour dietary recall, complete a physical activity questionnaire, and fill out a quality-of-life questionnaire. Additionally, anthropometric measurements and body composition analysis will be conducted. Blood samples will be collected to determine various biochemical parameters in the blood, including lipid profile (total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides), liver function tests, glucose, insulin, creatinine, urea, oxidative stress markers, inflammatory markers (C-reactive protein and lipopolysaccharides), and iron status markers. Furthermore, stool samples will be collected to analyze the composition of the intestinal microbiota and metabolomics.

To assess treatment adherence, participants will be provided with a food logs to record their daily food consumption during the initial visit. The participants will also receive a pantry containing protein-rich foods every week to facilitate the nutritional intervention. Also, 2 phone calls will be made each week to evaluate adherence to treatment. The adherence will be determined with the % of adherence to the dietary treatment as obtained in the analysis of the food logs.

ELIGIBILITY:
Inclusion Criteria:

Phase 1

* Signing of the informed consent form
* Both sexes
* Adults over 18 years of age
* BMI of 18.5 and under 40 kg/m2

Phase 2

* Both sexes
* Adults older than 18 years
* People with obesity (BMI of 30 to 40 kg/m2) and serum iron < 50 micrograms/dL.
* Total cholesterol less than 240 mg/dL (with the diet plan 20% decrease).

Exclusion Criteria:

* Any type of diabetes.
* Patients with renal disease diagnosed by a physician.
* Patients with acquired diseases that secondarily produce obesity and diabetes.
* Patients who have suffered a cardiovascular event.
* Weight loss > 3 kg in the last 3 months.
* Patients with catabolic diseases such as cancer and acquired immunodeficiency syndrome.
* Pregnancy.
* Treatment with any drug treatment:

  1. Treatment with antihypertensive drugs (loop or potassium-sparing diuretics, angiotensin-converting enzyme inhibitors (ACE inhibitors), angiotensin II receptor blockers, alpha blockers, calcium antagonists, beta blockers).
  2. Treatment with hypoglycemic agents (sulfonylureas, biguanides, incretins) or insulin and antidiabetics.
  3. Treatment with statins, fibrates or other drugs to control dyslipidemia.
  4. Use of steroid drugs, chemotherapy, immunosuppressants or radiotherapy.
  5. Anorectics or drugs that accelerate weight loss.
  6. Any drug or medication that activates intestinal motility (cisapride, dimethicone, domperidone, metoclopramide, trimebutine).
  7. Laxatives or antispasmodics 4 weeks prior to the study h) Antibiotic treatment 2 months prior to the study.
* Patients who have suffered a blood loss of more than 500 ml or recent gastrointestinal tract perforation.
* Patients with a smoking index greater than 21.
* Consumption of large amounts of alcohol (14 drinks for women or 21 drinks for men in a normal week).
* Consumption of any recreational psychoactive substance.
* Treatment with any medication that influences inflammation or iron metabolism (proton pump inhibitors, antacids, bisphosphonates, bile acid or calcium sequestrants).
* Patients who are vegetarians
* Allergy or intolerance to any food mentioned in the proposed pantry such as egg, dairy, fish, tuna, chicken, beans, lima beans and/or lentils.
* Unwillingness to consume any of the foods listed in the proposed pantry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
Serum hepcidin concentration in mcg/dL | Baseline to 2 months of intervention
  Change in serum hepcidin concentration between different nutritional interventions in subjects with obesity and iron deficiency

SECONDARY OUTCOMES:
Serum iron concentration in mcg/dL | Baseline to 2 months of intervention
  Change in serum iron concentration between different nutritional interventions in subjects with obesity and iron deficiency
Serum ferritin concentration in ng/mL | Baseline to 2 months of intervention
  Change in serum ferritin concentration between different nutritional interventions in subjects with obesity and iron deficiency
Serum iron binding capacity concentration in mcg/dL | Baseline to 2 months of intervention
  Change in serum iron binding capacity concentration between different nutritional interventions in subjects with obesity and iron deficiency
Blood reticulocytes percentage | Baseline to 2 months of intervention
  Change in blood reticulocytes percentage between different nutritional interventions in subjects with obesity and iron deficiency
Serum soluble transferrin receptor concentration in mg/L. | Baseline to 2 months of intervention
  Change in serum soluble transferrin receptor concentration between different nutritional interventions in subjects with obesity and iron deficiency
Blood haemoglobin concentration in g/dL | Baseline to 2 months of intervention
  Change in blood haemoglobin concentration between different nutritional interventions in subjects with obesity and iron deficiency
Serum C-reactive protein concentration in g/dL | Baseline to 2 months of intervention
  Change in C-reactive protein concentration between different nutritional interventions in subjects with obesity and iron deficiency
Serum leptin concentration in ng/mL | Baseline to 2 months of intervention
  Change in leptin concentration in the serum determined by ELISA kit between different nutritional interventions in subjects with obesity and iron deficiency
Serum interleukin 6 concentration in pg/mL | Baseline to 2 months of intervention
  Change in interleukin-6 concentration determined by ELISA kit between different nutritional interventions in subjects with obesity and iron deficiency
Serum lipopolysaccharides concentration in ng/mL | Baseline to 2 months of intervention
  Change in lipopolysaccharides concentration between different nutritional interventions in subjects with obesity and iron deficiency
Plasma malondialdehyde concentration in nmol/mL | Baseline to 2 months of intervention
  Change in malondialdehyde concentration by spectrophotometry between different nutritional interventions in subjects with obesity and iron deficiency
Plasma trolox equivalents concentration in umols/mL | Baseline to 2 months of intervention
  Change in trolox equivalents concentration between different nutritional interventions in subjects with obesity and iron deficiency
Changes in faecal microbiota composition | Baseline to 2 months of intervention
  The change in faecal microbiota composition shall be measured by 16 ribosome sequencing at baseline and at 2 months. The relative change of each bacterial taxon shall be calculated on the basis of the abundance of the given bacteria at baseline to 2 months between different nutritional interventions in subjects with obesity and iron deficiency
Serum total cholesterol concentration in mg/dL | Baseline to 2 months of intervention
  Change in total cholesterol concentration determined by autoanalyzer between different nutritional interventions in subjects with obesity and iron deficiency
Serum LDL cholesterol concentration in mg/dL | Baseline to 2 months of intervention
  Change in LDL-cholesterol concentration determined by autoanalyzer between different nutritional interventions in subjects with obesity and iron deficiency
Serum triglycerides concentration in mg/dL | Baseline to 2 months of intervention
  Change in triglycerides concentration determined by autoanalyzer between different nutritional interventions in subjects with obesity and iron deficiency
Serum aspartate aminotransferase concentration in IU/mL | Baseline to 2 months of intervention
  Change in aspartate aminotransferase concentration determined by autoanalyzer between different nutritional interventions in subjects with obesity and iron deficiency
Serum alanine aminotransferase concentration in IU/mL | Baseline to 2 months of intervention
  Change in alanine aminotransferase concentration determined by autoanalyzer between different nutritional interventions in subjects with obesity and iron deficiency
Serum glucose concentration in mg/dL | Baseline to 2 months of intervention
  Change in serum glucose concentration determined by autoanalyzer between different nutritional interventions in subjects with obesity and iron deficiency
Body weight in kilograms | Baseline to 2 months of intervention
  Change in body weight between different nutritional interventions in subjects with obesity and iron deficiency
Fat mass percentage | Baseline to 2 months of intervention
  Change in fat mass percentage determined by multifrequency electrical bioimpedance between different nutritional interventions in subjects with obesity and iron deficiency
Waist circumference in centimeters | Baseline to 2 months of intervention
  Change in waist circumference between different nutritional interventions in subjects with obesity and iron deficiency
Lean mass percentage | Baseline to 2 months of intervention
  Change in fat mass percentage determined by multifrequency electrical bioimpedance between different nutritional interventions in subjects with obesity and iron deficiency
Skeletal muscle mass percentage | Baseline to 2 months of intervention
  Change in fat mass percentage determined by multifrequency electrical bioimpedance between different nutritional interventions in subjects with obesity and iron deficiency

CONTACTS AND LOCATIONS:
Overall Officials: Martha Guevara-Cruz, MD, PhD, Principal Investigator — Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, México, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou Z, Zhang H, Chen K, Liu C. Iron status and obesity-related traits: A two-sample bidirectional Mendelian randomization study. Front Endocrinol (Lausanne). 2023 Feb 14;14:985338. doi: 10.3389/fendo.2023.985338. eCollection 2023. PMID 36864839
- [Background] Yanoff LB, Menzie CM, Denkinger B, Sebring NG, McHugh T, Remaley AT, Yanovski JA. Inflammation and iron deficiency in the hypoferremia of obesity. Int J Obes (Lond). 2007 Sep;31(9):1412-9. doi: 10.1038/sj.ijo.0803625. Epub 2007 Apr 17. PMID 17438557
- [Background] Becker C, Schumann K. Iron-homeostasis and obesity. J Trace Elem Med Biol. 2015 Apr;30:194. doi: 10.1016/j.jtemb.2014.06.009. Epub 2014 Jun 27. No abstract available. PMID 25023846
- [Background] Coimbra S, Catarino C, Santos-Silva A. The role of adipocytes in the modulation of iron metabolism in obesity. Obes Rev. 2013 Oct;14(10):771-9. doi: 10.1111/obr.12057. Epub 2013 Jul 11. PMID 23841713
- [Background] Collins JF, Wessling-Resnick M, Knutson MD. Hepcidin regulation of iron transport. J Nutr. 2008 Nov;138(11):2284-8. doi: 10.3945/jn.108.096347. PMID 18936232
- [Background] Anderson GJ, Frazer DM. Current understanding of iron homeostasis. Am J Clin Nutr. 2017 Dec;106(Suppl 6):1559S-1566S. doi: 10.3945/ajcn.117.155804. Epub 2017 Oct 25. PMID 29070551
- [Background] Ross AC. Impact of chronic and acute inflammation on extra- and intracellular iron homeostasis. Am J Clin Nutr. 2017 Dec;106(Suppl 6):1581S-1587S. doi: 10.3945/ajcn.117.155838. Epub 2017 Oct 25. PMID 29070546
- [Background] Joffin N, Gliniak CM, Funcke JB, Paschoal VA, Crewe C, Chen S, Gordillo R, Kusminski CM, Oh DY, Geldenhuys WJ, Scherer PE. Adipose tissue macrophages exert systemic metabolic control by manipulating local iron concentrations. Nat Metab. 2022 Nov;4(11):1474-1494. doi: 10.1038/s42255-022-00664-z. Epub 2022 Nov 3. PMID 36329217
- [Background] Gabrielsen JS, Gao Y, Simcox JA, Huang J, Thorup D, Jones D, Cooksey RC, Gabrielsen D, Adams TD, Hunt SC, Hopkins PN, Cefalu WT, McClain DA. Adipocyte iron regulates adiponectin and insulin sensitivity. J Clin Invest. 2012 Oct;122(10):3529-40. doi: 10.1172/JCI44421. Epub 2012 Sep 10. PMID 22996660
- [Background] Moreto F, de Oliveira EP, Manda RM, Burini RC. The higher plasma malondialdehyde concentrations are determined by metabolic syndrome-related glucolipotoxicity. Oxid Med Cell Longev. 2014;2014:505368. doi: 10.1155/2014/505368. Epub 2014 Jun 24. PMID 25089170
- [Background] Nikonorov AA, Skalnaya MG, Tinkov AA, Skalny AV. Mutual interaction between iron homeostasis and obesity pathogenesis. J Trace Elem Med Biol. 2015 Apr;30:207-14. doi: 10.1016/j.jtemb.2014.05.005. Epub 2014 May 24. PMID 24916791
- [Background] Teng IC, Tseng SH, Aulia B, Shih CK, Bai CH, Chang JS. Can diet-induced weight loss improve iron homoeostasis in patients with obesity: A systematic review and meta-analysis. Obes Rev. 2020 Dec;21(12):e13080. doi: 10.1111/obr.13080. Epub 2020 Jul 16. PMID 32677171
- [Background] Abbaspour N, Hurrell R, Kelishadi R. Review on iron and its importance for human health. J Res Med Sci. 2014 Feb;19(2):164-74. PMID 24778671
- [Background] Dev S, Babitt JL. Overview of iron metabolism in health and disease. Hemodial Int. 2017 Jun;21 Suppl 1(Suppl 1):S6-S20. doi: 10.1111/hdi.12542. Epub 2017 Mar 15. PMID 28296010
- [Background] Zhang C, Rawal S. Dietary iron intake, iron status, and gestational diabetes. Am J Clin Nutr. 2017 Dec;106(Suppl 6):1672S-1680S. doi: 10.3945/ajcn.117.156034. Epub 2017 Oct 25. PMID 29070554
- [Background] Frazer DM, Wilkins SJ, Becker EM, Vulpe CD, McKie AT, Trinder D, Anderson GJ. Hepcidin expression inversely correlates with the expression of duodenal iron transporters and iron absorption in rats. Gastroenterology. 2002 Sep;123(3):835-44. doi: 10.1053/gast.2002.35353. PMID 12198710
- [Background] Cao C, Thomas CE, Insogna KL, O'Brien KO. Duodenal absorption and tissue utilization of dietary heme and nonheme iron differ in rats. J Nutr. 2014 Nov;144(11):1710-7. doi: 10.3945/jn.114.197939. Epub 2014 Sep 10. PMID 25332470
- [Background] Chiabrando D, Vinchi F, Fiorito V, Mercurio S, Tolosano E. Heme in pathophysiology: a matter of scavenging, metabolism and trafficking across cell membranes. Front Pharmacol. 2014 Apr 8;5:61. doi: 10.3389/fphar.2014.00061. eCollection 2014. PMID 24782769
- [Background] Vela D. Hepcidin, an emerging and important player in brain iron homeostasis. J Transl Med. 2018 Feb 7;16(1):25. doi: 10.1186/s12967-018-1399-5. PMID 29415739
- [Background] Amato MC, Giordano C. Visceral adiposity index: an indicator of adipose tissue dysfunction. Int J Endocrinol. 2014;2014:730827. doi: 10.1155/2014/730827. Epub 2014 Apr 14. PMID 24829577
- [Background] Utami FA , Lee HC , Su CT , Guo YR , Tung YT , Huang SY . Effects of calorie restriction plus fish oil supplementation on abnormal metabolic characteristics and the iron status of middle-aged obese women. Food Funct. 2018 Feb 21;9(2):1152-1162. doi: 10.1039/c7fo01787a. PMID 29362766
- [Background] Mejia-Rodriguez F, Villalpando S, Shamah-Levy T, Garcia-Guerra A, Mendez-Gomez Humaran I, De la Cruz-Gongora VV. Prevalence of iron deficiency was stable and anemia increased during 12 years (2006-2018) in Mexican women 20-49 years of age. Salud Publica Mex. 2021 May 3;63(3 May-Jun):401-411. doi: 10.21149/12152. Spanish. PMID 34098613